CLINICAL TRIAL: NCT00000631
Title: A Phase I Randomized Trial to Evaluate the Safety and Immunogenicity of Vaccinia-HIV Envelope Recombinant Vaccine (HIVAC-1e) in Combination With Soluble Recombinant Envelope Vaccine (VaxSyn)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Prevention
Other Study IDs: AVEG 002B; 10539 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Envelope Proteins; Viral Vaccines; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia | interventions — HIVAC-1e; VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: HIVAC-1e
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
Primary: To determine whether additional boosting with soluble recombinant gp160 vaccine (VaxSyn) after priming with a vaccinia-HIV envelope recombinant (HIVAC-1e) provides a significant advantage in the degree and duration of immunogenicity. Secondary: To learn more about the safety of the combination use of the two HIV envelope vaccines in the study (VaxSyn and HIVAC-1e).

Recent Phase I trials conducted at the AIDS Vaccine Units have shown that antibodies have persisted in most recipients for 6 months after boosting, and responses seem significantly higher and more persistent than responses achieved by just two doses of soluble protein vaccine alone or two doses of HIVAC-1e alone. This study tests in a previously recruited cohort of volunteers whether additional boosting with soluble recombinant gp160 results in increased immunogenicity of longer duration.

DETAILED DESCRIPTION:
Recent Phase I trials conducted at the AIDS Vaccine Units have shown that antibodies have persisted in most recipients for 6 months after boosting, and responses seem significantly higher and more persistent than responses achieved by just two doses of soluble protein vaccine alone or two doses of HIVAC-1e alone. This study tests in a previously recruited cohort of volunteers whether additional boosting with soluble recombinant gp160 results in increased immunogenicity of longer duration.

Twelve volunteers who have previously received two doses of HIVAC-1e (or DryVax) and two doses of gp160 receive an additional boost of gp160 at 12-20 months after the last boost and an additional dose of HIVAC-1e at least 9 months after the final gp160 boost.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Normal history and physical exam.
* Negative ELISA for HIV.
* Negative HIV p24 antigen test.
* Normal urinalysis.

Prior Medication: Required:

* Two prior doses of HIVAC-1e (or DryVax) and two prior doses of gp160 vaccine.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Risk factors for HIV infection including active intravenous drug use and more than 2 sexual partners.
* History of immunodeficiency or chronic illness.
* Hypersensitivity to insects.
* Medical or psychiatric condition that makes it unlikely the patient will comply with the protocol.

Patients with the following prior conditions are excluded:

* History of immunodeficiency or chronic illness.

Prior Medication:

Excluded:

* Immunosuppressive medications.

Prior Treatment:

Excluded:

* Blood or blood product transfusion within the past 6 months.

Risk Behavior: Excluded:

* Intravenous drug use.
* More than 2 sexual partners.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13
Dates: Study Completion 1992-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey L, Study Chair
Locations (1):
- Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington, United States

REFERENCES:
- [Background] McElrath MJ, Corey L, Greenberg PD. Evaluation of cytotoxic T cell responses to candidate HIV-1 vaccines in HIV-1-uninfected individuals. AIDS Res Hum Retroviruses. 1994;10 Suppl 2:S69-72. PMID 7865336
- [Background] Kent SJ, Greenberg PD, Hoffman MC, Akridge RE, McElrath MJ. Antagonism of vaccine-induced HIV-1-specific CD4+ T cells by primary HIV-1 infection: potential mechanism of vaccine failure. J Immunol. 1997 Jan 15;158(2):807-15. PMID 8992998
- [Background] Mosier DE, Gulizia RJ, MacIsaac PD, Corey L, Greenberg PD. Resistance to human immunodeficiency virus 1 infection of SCID mice reconstituted with peripheral blood leukocytes from donors vaccinated with vaccinia gp160 and recombinant gp160. Proc Natl Acad Sci U S A. 1993 Mar 15;90(6):2443-7. doi: 10.1073/pnas.90.6.2443. PMID 8460155
- [Background] McElrath J, Peterson E, Dragavon J, Berger D, Hoffman M, Klucking S, Greenberg P, Corey L. Combination prime-boost approach to HIV vaccination in seronegative individuals: enhanced immunity with additional subunit gp160 protein boosting. Int Conf AIDS. 1992 Jul 19-24;8(1):Mo9 (abstract no MoB 0027)
- [Background] McElrath MJ, Rabin M, Hoffman M, Klucking S, Garcia JV, Greenberg PD. Evaluation of human immunodeficiency virus type 1 (HIV-1)-specific cytotoxic T-lymphocyte responses utilizing B-lymphoblastoid cell lines transduced with the CD4 gene and infected with HIV-1. J Virol. 1994 Aug;68(8):5074-83. doi: 10.1128/JVI.68.8.5074-5083.1994. PMID 8035507
- [Background] McElrath MJ, Corey L, Greenberg PD, Matthews TJ, Montefiori DC, Rowen L, Hood L, Mullins JI. Human immunodeficiency virus type 1 infection despite prior immunization with a recombinant envelope vaccine regimen. Proc Natl Acad Sci U S A. 1996 Apr 30;93(9):3972-7. doi: 10.1073/pnas.93.9.3972. PMID 8633000
- [Background] Cooney EL, McElrath MJ, Corey L, Hu SL, Collier AC, Arditti D, Hoffman M, Coombs RW, Smith GE, Greenberg PD. Enhanced immunity to human immunodeficiency virus (HIV) envelope elicited by a combined vaccine regimen consisting of priming with a vaccinia recombinant expressing HIV envelope and boosting with gp160 protein. Proc Natl Acad Sci U S A. 1993 Mar 1;90(5):1882-6. doi: 10.1073/pnas.90.5.1882. PMID 8446603